CLINICAL TRIAL: NCT02906774
Title: A Prospective, Case-series Study of Fecal Microbiota Transplantation for the Selective Intestinal Decolonization of Multidrug-resistant, Pathogenic Enterobacteriaceae
Brief Title: Fecal Transplant for MDR Pathogen Decolonization
Status: Terminated | Type: Observational
Why Stopped: This observational study has been transitioned to a clinical trial and is now registered at (NCT04181112).
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Amee Manges, Associate Professor, University of British Columbia
Other Study IDs: H15-01944
Record Dates: First submitted 2016-08-08; First posted 2016-09-20 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Multi-antibiotic Resistance
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool specimens from FMT donors and recipients.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Fecal microbiota transplantation (FMT) — Fecal microbiota transplantation after antibiotic pretreatment

SUMMARY:
This is a proof-of-principle research study designed to determine whether fecal microbiota transplantation (FMT) can eliminate highly drug-resistant bacteria from the intestinal tract of renal transplant patients. The primary goal of this study is to test whether oral gut decontamination followed by FMT by enema delivery will result in decolonization of the intestinal tract of renal transplant patients shortly after solid organ transplantation, thereby preventing difficult to treat post-transplant infections.

DETAILED DESCRIPTION:
Contact the study principal investigator for the study protocol.

ELIGIBILITY:
Renal transplant patient inclusion criteria:

* 18 years or older
* Able to provide informed consent
* Positive for one of the target MDR organisms by rectal or stool culture tests

FMT stool donor inclusion criteria:

* Able to provide informed consent
* Able to complete donor screening
* Able to adhere to FMT stool collection and testing procedures

Renal transplant patient exclusion criteria:

* Still in hospital at week 7 following organ transplantation
* Pregnant or planning to become pregnant
* Breastfeeding
* Participating in another interventional or investigational study
* Neutropenic (ANC < 0.5)
* Colonized with Clostridium difficile
* Presence of colostomy or ileostomy
* Has an active intestinal infection
* Fever > 38.0 or WBC count > 15,000
* Are taking a non-dietary probiotic supplement
* Require or are expected to require systemic antimicrobial therapy other than Pneumocystis prophylaxis or cytomegalovirus (CMV) therapy during the study period
* Has a severe underlying disease with anticipated survival less than 6 months
* Are unable to tolerate FMT or enema for any reason, or where their physician believes for any reason that FMT might pose a health risk to the subject
* Subjects who report a history of anaphylactoid food allergy will not be excluded but these allergies will be noted and donors will be required to avoid ingestion of these foods for at least three days prior to donation

FMT stool donor exclusion criteria:

* Presence of any of the following by stool examination: vancomycin-resistant Enterococci (VRE), Salmonella, Shigella, shiga toxin-producing E. coli, Yersinia, Campylobacter, ESBL or carbapenemase-producing Enterobacteriaceae (CRE), pathogenic ova or parasites, C. difficile toxin B (by PCR), or rotavirus, adenovirus and norovirus
* History of any type of active cancer aside from melanoma
* Risk factors for acquisition of HIV, syphilis, Hepatitis B, Hepatitis C, prion or any neurological disease as determined by the donor questionnaire
* History of gastrointestinal comorbidities, e.g., inflammatory bowel disease, irritable bowel syndrome, chronic constipation or diarrhea, or colostomy or ileostomy
* Receipt of blood transfusion from a country other than Canada in the preceding 6 months
* Antibiotic use or any systemic immunosuppressive agents in the 3 months prior to stool donation
* Receipt of any live vaccine within 3 months prior to stool donation
* Any current or previous medical or psychosocial condition or behaviors which in the opinion of the investigator may pose risk to the recipients or the donor

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant patients who are intestinally colonized with any of the target MDR organisms based on rectal culture screening according to Provincial Infection Control Network of British Columbia guidelines and performed by the Vancouver General Hospital Clinical Laboratory will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study will be the proportion of successfully decolonized patients out of all study patients evaluated, defined as the sustained elimination of a MDR target organism over a minimum of ≥ 2 study visits. | 6 months

SECONDARY OUTCOMES:
Determine the number of patients with treatment-related adverse events, as defined by the study adverse event questionnaire (including the Common Terminology Criteria for Adverse Events (v4.0)). | 6 months
Estimate the proportion of patients who become re-colonized following FMT. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amee Manges, MPH, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided